CLINICAL TRIAL: NCT04527367
Title: Epidemiology and Long-term Prognosis of Patients With Valvular Heart Diseases (BIA-WAD Study)
Brief Title: Epidemiology and Long-term Outcome of Patients With VHD
Acronym: BIA-WAD
Status: Completed | Type: Observational
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Principal Investigator, Lukasz Kuzma, Principal Investigator,, Medical University of Bialystok
Other Study IDs: UMB-KKI-101
Record Dates: First submitted 2020-08-22; First posted 2020-08-26 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: Valvular Disease; Valvular Heart Disease; Aortic Valve Stenosis; Mitral Insufficiency and Aortic Stenosis; Mitral Stenosis; Coronary Artery Disease; Chronic Kidney Diseases
Keywords: Valvular Heart Disease; Aortic Valve Stenosis; Mitral Insufficiency; Coronary Artery Disease; Chronic Kidney Diseases
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Stenosis; Mitral Valve Insufficiency; Mitral Valve Stenosis; Coronary Artery Disease; Renal Insufficiency, Chronic | interventions — Cardiac Surgical Procedures; Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VHD patients: Patients with moderate and severe valvular heart diseases
  Interventions: Procedure: Innovative medical technologies in invasive cardiology and cardiac surgery

INTERVENTIONS:
Procedure: Innovative medical technologies in invasive cardiology and cardiac surgery — A follow-up study included the analysis of medical documentation of the Cardiosurgery and the Invasive Cardiology Departments to provided information on the duration and type of procedure performed.
  Other Names: Percutaneous coronary intervention; Percutaneous aortic valve replacement; Percutaneous interventional mitral regurgitation treatment; Cardiosurgery

SUMMARY:
Valvular heart diseases are significant problem in Polish population. Coexistence of coronary artery disease in patients with VHD increases the risk of death and affects further therapeutic strategy. The aim of the study is analysis the epidemiology and the long-term prognosis among patients with VHD.

DETAILED DESCRIPTION:
Valvular heart diseases are significant problem in Polish population. Coexistence of coronary artery disease in patients with VHD increases the risk of death and affects further therapeutic strategy.

Patients with moderate and severe valvular heart diseases are included into the study. The set of variables subject to interpretation consisted of demographic data, medical history, result of coronary angiography, and type of applied percutaneous and surgical treatment

ELIGIBILITY:
Inclusion Criteria:

* Valvular heart disease in moderate and severe stages

Exclusion Criteria:

* Age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in Medical University of Bialystok.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Death | 3665 days
  All-cause of mortality

SECONDARY OUTCOMES:
MACCE | 3665 days
  Mocardial infarction, stent thrombosis, stroke or transient ischemic attack, urgent revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Łukasz Kuźma, MD, PhD, Principal Investigator — Medical University of Bialystok
Locations (1):
- Department of Invasive Cardiology, Medical University of Bialystok, The Medical University of Bialystok Clinical Hospital, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kuzma L, Bachorzewska-Gajewska H, Kozuch M, Struniawski K, Pogorzelski S, Hirnle T, Dobrzycki S. Acute coronary syndromes and atherosclerotic plaque burden distribution in coronary arteries among patients with valvular heart disease (BIA-WAD registry). Postepy Kardiol Interwencyjnej. 2019;15(4):422-430. doi: 10.5114/aic.2019.90216. Epub 2019 Dec 8. PMID 31933658
- [Result] Kuzma L, Malyszko J, Bachorzewska-Gajewska H, Niwinska MM, Kurasz A, Zalewska-Adamiec M, Kozuch M, Dobrzycki S. Impact of chronic kidney disease on long-term outcome of patients with valvular heart defects. Int Urol Nephrol. 2020 Nov;52(11):2161-2170. doi: 10.1007/s11255-020-02561-4. Epub 2020 Jul 14. PMID 32661631